CLINICAL TRIAL: NCT02575924
Title: Employing a Single Step Media Can Improve the Clinical Outcomes in Those Patient Who Usually Show an High Cycle Cancellation Rate?
Brief Title: Influence of Culture Media on Clinical Outcomes in Poor Responders or Severe Male Infertility
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MGM13
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Poor Responder; Severe Male Infertility; Embryo Development; Blastocyst; Culture Media
Keywords: media; blastocyst; male infertility; poor responders; pgs
MeSH Terms: conditions — Infertility, Male; Mental Retardation, X-Linked 59

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- sequential medium female age>=40 (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE-FERT medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE-CLEAVAGE medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day3
  day3: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices and newer volumes of mineral oil to cover up the droplets till day5
  day5: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices without any mineral oil replacement till day7
  Interventions: Drug: sequential medium
- sequential medium female age<40 (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE-FERT medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE-CLEAVAGE medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day3
  day3: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices and newer volumes of mineral oil to cover up the droplets till day5
  day5: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices without any mineral oil replacement till day7
  Interventions: Drug: sequential medium
- sequential medium sperm testis retrieval (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE-FERT medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE-CLEAVAGE medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day3
  day3: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices and newer volumes of mineral oil to cover up the droplets till day5
  day5: fitting volumes of SAGE-BLASTOCYSTS medium to replace all the culture devices without any mineral oil replacement till day7
  Interventions: Drug: sequential medium
- one step medium female age>=40 (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE 1-STEP medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE 1-STEP medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day7
  Interventions: Drug: 1-step medium
- one step medium female age<40 (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE 1-STEP medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE 1-STEP medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day7
  Interventions: Drug: 1-step medium
- one step medium sperm testis retrieval (Active Comparator): day 0: suitable number of test tubes, each one filled with 1ml of SAGE 1-STEP medium to gather all the oocytes retrieved during the pick up (at most 3 oocytes/test tube)
  1 or more culture dish with 6 droplets (35µl) of SAGE 1-STEP medium covered with mineral oil to culture the zygotes/embryos after ICSI procedure till day7
  Interventions: Drug: 1-step medium

INTERVENTIONS:
Drug: sequential medium — administration of Quinn's Advantage® Fertilization Medium on day0 administration of Quinn's Advantage® Cleavage Medium from day0 to day3 administration of Quinn's Advantage® Blastocyst Medium from day3 to day7
  Other Names: Quinn's Advantage® Fertilization Medium; Quinn's Advantage® Cleavage Medium; Quinn's Advantage® Blastocyst Medium
  Arms: sequential medium female age<40; sequential medium female age>=40; sequential medium sperm testis retrieval
Drug: 1-step medium — administration of SAGE 1-Step™ with Human Albumin Solution, from day0 to day7
  Other Names: SAGE 1-Step™ with Human Albumin Solution
  Arms: one step medium female age<40; one step medium female age>=40; one step medium sperm testis retrieval

SUMMARY:
In this study the suitability of two -sequential and single step- commercially available culture media from the same brand was compared. The aim of such study is to verify whether is possible to improve the efficiency of infertility treatments in those couples who usually have a high cycle cancellation rate, such as poor responder patients and severe male infertility. The study population is composed of couples attending the fertility clinic: to this purpose all those couples approaching IVF treatments with a diagnosis of OAT, cryptozoospermia, advanced maternal age and women with a "poor responder" diagnosis were recruited. IVF treatments were randomly set to be cultured either with two-step sequential media or with one-step media to acquire data concerning the ongoing embryo culture development and clinical outcomes.

DETAILED DESCRIPTION:
The final goal in the field of Assisted Reproductive Technology is to obtain a single healthy newborn. For that purpose, a lot of factors are strictly interconnected each other's and have to be carefully evaluated. The choice of embryo culture system and of embryo selection strategy plays a crucial role in obtain and identify the embryo with the highest implantation potential. One really important key factor is the choice of the culture media. Currently, there are numerous commercially available culture media showing very different compositions. Essentially two strategies have been applied for the design of culture media: 1) "Back to nature" for sequential media, based on the physiology of the embryo and the measured concentration of substances present in its natural environment and 2) "Let the embryo choose" for single step media, where none a priori assumption of the concentration of a component is made. In the literature, there are a lot of studies analyzing the effect of culture media on human preimplantation embryos development and comparing biological and clinical outcomes among different media compositions. Several studies performed a comparison about the development of human zygotes in either a one-step or two-step culture system. Usually there were no significant differences between the two culture media systems regarding biological or clinical outcomes. Anyway, a greater number of blastocysts were generally obtained by the continuous single medium culture if compared with sequential culture media, even if the implantation and clinical pregnancy rates are comparable.

ELIGIBILITY:
Inclusion Criteria:

* advanced maternal age,
* poor responder women (<=4 oocytes),
* cryptozoospermia,
* testicular retrieval of spermatozoa

Exclusion Criteria:

* any other

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
blastocystis development rate | six months
implantation rate | six months
clinical pregnancy rate | one year
  total number of gestational chambers resulting from the total embryo transferred

SECONDARY OUTCOMES:
ploidy status | six months
  Embryo genetic status after chromosomal screening

CONTACTS AND LOCATIONS:
Overall Officials: MariaGiulia Minasi, Biology, Principal Investigator — European Hospital
Locations (1):
- Center for Reproductive Medicine, Rome, RM, Italy

REFERENCES:
- [Background] Basile N, Morbeck D, Garcia-Velasco J, Bronet F, Meseguer M. Type of culture media does not affect embryo kinetics: a time-lapse analysis of sibling oocytes. Hum Reprod. 2013 Mar;28(3):634-41. doi: 10.1093/humrep/des462. Epub 2013 Jan 12. PMID 23315059
- [Background] Biggers JD, Summers MC. Choosing a culture medium: making informed choices. Fertil Steril. 2008 Sep;90(3):473-83. doi: 10.1016/j.fertnstert.2008.08.010. PMID 18847602
- [Background] Chronopoulou E, Harper JC. IVF culture media: past, present and future. Hum Reprod Update. 2015 Jan-Feb;21(1):39-55. doi: 10.1093/humupd/dmu040. Epub 2014 Jul 17. PMID 25035437
- [Background] Ciray HN, Aksoy T, Goktas C, Ozturk B, Bahceci M. Time-lapse evaluation of human embryo development in single versus sequential culture media--a sibling oocyte study. J Assist Reprod Genet. 2012 Sep;29(9):891-900. doi: 10.1007/s10815-012-9818-7. Epub 2012 Jun 20. PMID 22714134
- [Background] Gardner DK, Lane M. One-step versus two-step culture of mouse preimplantation embryos. Hum Reprod. 2006 Jul;21(7):1935-6; author reply 1936-9. doi: 10.1093/humrep/del070. No abstract available. PMID 16818962
- [Background] Lane M, Gardner DK. Embryo culture medium: which is the best? Best Pract Res Clin Obstet Gynaecol. 2007 Feb;21(1):83-100. doi: 10.1016/j.bpobgyn.2006.09.009. Epub 2006 Nov 7. PMID 17090393
- [Background] Mantikou E, Youssef MA, van Wely M, van der Veen F, Al-Inany HG, Repping S, Mastenbroek S. Embryo culture media and IVF/ICSI success rates: a systematic review. Hum Reprod Update. 2013 May-Jun;19(3):210-20. doi: 10.1093/humupd/dms061. Epub 2013 Feb 5. PMID 23385469
- [Background] Reed ML, Hamic A, Thompson DJ, Caperton CL. Continuous uninterrupted single medium culture without medium renewal versus sequential media culture: a sibling embryo study. Fertil Steril. 2009 Nov;92(5):1783-6. doi: 10.1016/j.fertnstert.2009.05.008. Epub 2009 Jun 12. PMID 19523617
- [Background] Summers MC, Bird S, Mirzai FM, Thornhill A, Biggers JD. Human preimplantation embryo development in vitro: a morphological assessment of sibling zygotes cultured in a single medium or in sequential media. Hum Fertil (Camb). 2013 Dec;16(4):278-85. doi: 10.3109/14647273.2013.806823. Epub 2013 Jul 17. PMID 23862646